CLINICAL TRIAL: NCT04745507
Title: Outreach Crisis Intervention With a Team-based and Integrative Model of Treatment (AKtiV Study): Evaluation of the Inpatient Equivalent HomeTreatment (IEHT According to the German Social Code Book §115d SGB V) - a Proof-of-Concept Study
Brief Title: Implementation, Efficacy and Costs of Inpatient Equivalent Home-Treatment in German Mental Health Care
Acronym: AKtiV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Vivantes Netzwerk für Gesundheit GmbH (Other)
Collaborators: Medizinische Hochschule Brandenburg Theodor Fontane (Other); Zentrum für Psychiatrie Südwürttemberg (Unknown); Isar-Amper Klinikum München Ost (Unknown); Klinik für Psychiatrie und Psychotherapie II der Universität Ulm (Unknown); Kompetenzzentrum für Klinische Studien, Bremen (Unknown); Vivantes Klinikum am Urban (Unknown)
Responsible Party: Principal Investigator, Sebastian von Peter, Prof. Dr. med. Sebastian von Peter, Medizinische Hochschule Brandenburg Theodor Fontane
Other Study IDs: 01VSF19048
Record Dates: First submitted 2021-01-07; First posted 2021-02-09 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Mental Disorder; Personality Disorders; Schizo Affective Disorder; Anxiety Disorders; Eating Disorders; Addiction
Keywords: community mental health care; inpatient-equivalent home treatment; crisis resolution teams
MeSH Terms: conditions — Mental Disorders; Personality Disorders; Psychotic Disorders; Anxiety Disorders; Feeding and Eating Disorders; Behavior, Addictive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Arm 1 / C1: This cohort (C1) consists of 180 patients who receive IEHT in the recruiting sites, fulfil inclusion criteria and gave informed consent regarding their study participation.
  Interventions: Other: Inpatient Equivalent Home Treatment
- Arm 2 / C2: This cohort (C2) consist of 180 patients receiving standard inpatient care (TAU) from the IEHT delivering hospital who fulfil inclusion criteria, are identified through a propensity score (PS) function as optimal control user or rather a "PS match" and gave informed consent regarding their study participation
- Arm 3: 360 close relatives or informal caregivers living in the same household of the participating patients who gave informed consent regarding their study participation. Thereby, one relative of each patients who is participating in the trial will be assessed (C1 = 180, C2 = 180).
- Arm 4:: Staff members of participating study cites as well as local and political stakeholders engaged with IEHT who gave informed consent (approximately n = 100 participants overall).

INTERVENTIONS:
Other: Inpatient Equivalent Home Treatment — At-home psychiatric treatment by means of a multiprofessional clinic team (an equivalent to stationary psychiatric care).
  Groups: Arm 1 / C1

SUMMARY:
The "inpatient-equivalent home treatment"(IEHT) according to §115d SGB-V is a particular version of the internationally well-known and evidence-based Home Treatment. As a complex intervention, IEHT requires a multi-method evaluation on different levels in the German context. The AKtiV study that is financed by the Innovation Fund of the Federal Joint Committee (proposal ID: VSF2_2019-108) meets this request. In this quasi-experimental study with a propensity score-matched control group, we assess and combine quantitative and qualitative data. Outcome parameters include classical clinical ones such as hospital readmission rates, mental state, and recovery outcomes. In addition, it evaluates issues concerning the right target population, treatment processes, implementation strategies, and factors associated with positive outcomes. The study takes into account the perspective of patients, relatives, staff as well as decision makers in politics and administration. Therefore, we expect the results to be relevant for a broad audience and to contribute to further refinement and adaption of the model.

DETAILED DESCRIPTION:
The overarching goal of the AKtiV trial is to examine implementation processes, treatment processes, clinical efficacy, costs, and subjective experiences of IEHT following §115d of the German Social Code Book Five (SGB-V)compared to inpatient treatment from the perspective of service users, relatives or rather informal care givers' , staff and other stakeholders in mental health care. To maximize transferability of study results and to cover a broad spectrum of IEHT experience, 10 hospitals from different regions of Germany (e.g. rural, urban, east, west) participate in this study. Combining routine data, primary data and prospective follow-up data, the study results will be based/ involve a comprehensive database. Further, the combination of clinical and health economic data will enable the assessment of costs and benefits from a national perspective, a particularity of importance, given that there are only a few studies with health economic evidence of acute outreach mental health care. The qualitative evaluation of processes and out-comes of IEHT uses a collaborative-participatory approach that aligns with current demands for more user orientation and/ or involvement of people and researchers with lived experience in the process of developing interventions and their evaluation. The mixed-methods design of the trial corresponds with current standards of empirical social research enabling the triangulation of hypothesis-confirming, quantifiable factors and hypothesis-generating, qualitative aspects. By parallelizing on one hand quantitative and qualitative data and on the other hand routine data with primary data, data on implementation processes and data on treatment processes, different facets from different perspectives and levels of IEHT are targeted. This allows for a comprehensive, holistic assessment of this innovative treatment offer.

ELIGIBILITY:
For C1 and C2:

Inclusion criteria:

* IEHT inclusion criteria

  * acute mental health crisis that requires inpatient treatment;
  * social and living surrounding allowing for home visits and private conversations;
  * informed consent of all adults living in the service user's place of residency;
* ability to provide informed consent
* sufficient German language skills
* permanent residence in the catchment area of the IEHT delivering Hospital
* main diagnosis within the ICD codes F0X, F1X, F2X, F3X, F4X, F5X, or F6X

Exclusion criteria:

* IEHT exclusion criteria

  o in case of children living in the same household, presence of child welfare risk
* acute suicidality or aggressiveness towards others requiring hospital admission
* Being under order of commitment
* participation in an interventional study during the recruitment
* presence of substantial cognitive deficits as indicated by severe organic brain disease
* diagnosis of intellectual impairment
* admission longer ago than 7 days

For C3: Close relative or informal caregiver living in the same household of the participating patient

Inclusion criteria:

• informed consent regarding study participation

For C4: IEHT staff member of participating study cite OR local or political stakeholder engaged with IEHT

Inclusion criteria:

• informed consent regarding study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: C1: This cohort consists of patients who receive IEHT in the recruiting sites.
  C2: This cohort consits of patients receiving standard inpatient care (treatment as usual / TAU) from the IEHT delivering hospital
  C3: This cohort consits of close relatives or informal caregivers living in the same househod of the participating patients.
  C4: Staff members of participatimg study cites as well as local and political stakeolders engaged with IEHT
Sampling Method: Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Differences and change in the hospital re-admission rate | (T0.1) within 7 days after admission, (T1) 6 months after T0.1, (T2) 12 months after T0.1
  Observed Differences and change in the hospital re-admission of service users (C1 and C2) within 12 months after inclusion into the trial assessed via routine data of the study sites and the German Version oft the Client Sociodemographic and Service Receipt Inventory (CSSR-D; Roick et al., 2001).

SECONDARY OUTCOMES:
Combined readmission (day clinic, IEHT or hospital) | (T0.1) within 7 days after admission, (T1) 6 months after T0.1, (T2) 12 months after T0.1
  Combined readmission (day clinic, IEHT or hospital) of service users (C1 and C2) within 12 months after inclusion into the trial assessed via routine data of the study sites and the German Version oft the Client Sociodemographic and Service Receipt Inventory (CSSR-D; Roick et al., 2001).
Continuity of care | [Time Frame: (T0.1) within 7 days after admission, (T0.2) 7 days before or after discharge , (T1) 6 months after T0.1, (T2) 12 months after T0.1]
  The amount of service users (C1 and C2) dropping out of treatment after inclusion into the trial assessed via routine data of the study sites and the German Version oft the Client Sociodemographic and Service Receipt Inventory (CSSR-D; Roick et al., 2001).
Total number of inpatient days | (T0.1) within 7 days after admission, (T1) 6 months after T0.1, (T2) 12 months after T0.1
  Total number of inpatient days of service users (C1 and C2) after inclusion into the trial assessed via routine data of the study sites and the German Version of the Client Sociodemographic and Service Receipt Inventory (CSSR-D; Roick et al., 2001).
Generic health status | (T0.1) within 7 days after admission, (T1) 6 months after T0.1, (T2) 12 months after T0.1
  Generic health status of service users (C1 and C2) after inclusion into the trial assessed via the German Version of the EQ-5D-5L (Ludwig, von der Schulenburg, & Greiner, 2017).
Psychosocial functioning | (T0.1) within 7 days after admission, (T1) 6 months after T0.1, (T2) 12 months after T0.1
  The psychosocial functioning of service users (C1 and C2) after inclusion into the trial assessed via the German Version of the Health of the Nation Outcome Scales (HoNOS-D; Andreas S. et. al., 2007).
  * the unabbreviated scale title: Health of the Nation Outcome Scales
  * the minimum and maximum values: 0, 48
  * higher scores mean a worse outcome.
Personal and Social functioning | (T0.1) within 7 days after admission, (T1) 6 months after T0.1, (T2) 12 months after T0.1
  The level Personal and Social functioning of service users (C1 and C2) after inclusion into the trial assessed via the German Version of the Personal and Social Performance Scale (PSP; Schaub & Juckel, 2011).
  * the unabbreviated scale title: Deutsche Version der Personal and Social Performance Scale
  * the minimum and maximum values: 0, 100
  * higher scores mean a better outcome.
Professional reintegration | (T0.1) within 7 days after admission, (T1) 6 months after T0.1, (T2) 12 months after T0.1
  The professional/work reintegration of service users (C1 and C2) after inclusion into the trial assessed via the German Version oft the Client Sociodemographic and Service Receipt Inventory (CSSR-D; Roick et al., 2001).
Personal Recovery | (T0.1) within 7 days after admission, (T1) 6 months after T0.1, (T2) 12 months after T0.1
  Personal recovery of service users (C1 and C2) after inclusion into the trial assessed via the German Version of the Recovery Assessment Scale (RAS-G; Cavelti et. al, 2016).
  * the unabbreviated scale title: Recovery Assessment Scale-German Version
  * the minimum and maximum values: 14, 70
  * higher scores mean a better outcome.
Cost-utility | (T0.1) within 7 days after admission, (T1) 6 months after T0.1, (T2) 12 months after T0.1
  Cost-utility including direct and indirect disease related costs of service users (C1 and C2) after inclusion into the trial assessed via the German Version oft the Client Sociodemographic and Service Receipt Inventory (CSSR-D; Roick et al., 2001).
Quality-adjusted life year | (T0.1) within 7 days after admission, (T1) 6 months after T0.1, (T2) 12 months after T0.1
  Quality-adjusted life years of service users (C1 and C2) after inclusion into the trial assessed via the German Version of the EQ-5D-5L (Ludwig, von der Schulenburg, & Greiner, 2017)
Treatment satisfaction | (T0.2) 7 days before or after discharge
  The treatment satisfaction of service users (C1 and C2) assessed by a self developed questionnaire.
  * the unabbreviated scale title: Behandlungszufriedenheit
  * the minimum and maximum values: 0, 72
  * higher scores mean a better outcome.
Treatment satisfaction of close relatives or informal caregiver | (T0.2) 7 days before or after discharge
  The treatment satisfaction of close relatives or informal caregiver (C3) for both groups (C1 and C2) assessed by a self developed questionnaire.
  * the unabbreviated scale title: Zufriedenheitsbefragung Angehörige
  * the minimum and maximum values: 0, 52
  * higher scores mean a better outcome.
Burden of close relatives or informal caregiver | (T0.2) 7 days before or after discharge
  Burden of close relatives or informal caregiver (C3) for both groups (C1 and C2) assessed by via the German Version of the Involvement Evaluation Questionnaire (IEQ-EU; Bernert, et. al, 2001).
  * the unabbreviated scale title: Involvement Evaluation Questionnaire
  * the minimum and maximum values: 0, 120
  * higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian von Peter, Prof. Dr., Study Director — Immanuel Klinik Rüdersdorf; Andreas Bechdolf, Prof. Dr., Principal Investigator — Vivantes Klinikum am Urban
Locations (10):
- Germany (10):
  - Zentrum für Psychiatrie Reichenau, Reichenau, Baden-Wurttemberg
  - PP.rt, Gemeinnützige Gesellschaft für Psychiatrie Reutlingen mbH,, Reutlingen, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Klinik für Psychiatrie und Psychotherapie, Tübingen, Baden-Wurttemberg
  - Klinik für Psychiatrie und Psychotherapie I der Universität Ulm (Weissenau),, Weißenau, Baden-Wurttemberg
  - • Zentrum für Psychiatrie Südwürttemberg, Klinik für Psychiatrie und Psychotherapie Zwiefalten, Zwiefalten, Baden-Wurttemberg
  - kbo-Isar-Amper-Klinikum München-Ost, Haar, Bavaria
  - Immanuel Klinik Rüdersdorf, Abteilung für Psychiatrie, Psychotherapie und Psychosomatik, Psychiatrische Hochschulklinik, Rüdersdorf, Brandenburg
  - Vivantes Klinikum am Urban; Klinik für Psychiatrie, Psychotherapie und Psychosomatik, Kreuzberg, State of Berlin
  - • Klinik für Psychiatrie und Psychotherapie, Campus Charité Mitte,, Mitte, State of Berlin
  - Vivantes Neukölln, Klinik für Psychiatrie, Psychotherapie und Psychosomatik, Berlin

REFERENCES:
- [Background] Roick C, Kilian R, Matschinger H, Bernert S, Mory C, Angermeyer MC. [German adaptation of the client sociodemographic and service receipt inventory - an instrument for the cost of mental health care]. Psychiatr Prax. 2001 Oct;28 Suppl 2:S84-90. doi: 10.1055/s-2001-17790. German. PMID 11605129
- [Background] Andreas S, Harfst T, Dirmaier J, Kawski S, Koch U, Schulz H. A Psychometric evaluation of the German version of the 'Health of the Nation Outcome Scales, HoNOS-D': on the feasibility and reliability of clinician-performed measurements of severity in patients with mental disorders. Psychopathology. 2007;40(2):116-25. doi: 10.1159/000098492. Epub 2007 Jan 11. PMID 17215598
- [Background] Cavelti M, Wirtz M, Corrigan P, Vauth R. Recovery assessment scale: Examining the factor structure of the German version (RAS-G) in people with schizophrenia spectrum disorders. Eur Psychiatry. 2017 Mar;41:60-67. doi: 10.1016/j.eurpsy.2016.10.006. Epub 2016 Dec 31. PMID 28049083
- [Background] Bernert S, Kilian R, Matschinger H, Mory C, Roick C, Angermeyer MC. [The assessment of burden on relatives of mentally ill people: the German version of the involvement evaluation questionnaire (IEQ-EU)]. Psychiatr Prax. 2001 Oct;28 Suppl 2:S97-101. doi: 10.1055/s-2001-17792. German. PMID 11605131
- [Background] Ludwig K, von der Schulenburg JG, Greiner W. Valuation of the EQ-5D-5L with composite time trade-off for the German population - an exploratory study. Health Qual Life Outcomes. 2017 Feb 20;15(1):39. doi: 10.1186/s12955-017-0617-9. PMID 28219389
- [Background] Schaub D, Juckel G. [PSP Scale: German version of the Personal and Social Performance Scale: valid instrument for the assessment of psychosocial functioning in the treatment of schizophrenia]. Nervenarzt. 2011 Sep;82(9):1178-84. doi: 10.1007/s00115-010-3204-4. German. PMID 21174069
- [Derived] Bechdolf A, Nikolaidis K, von Peter S, Langle G, Brieger P, Timm J, Killian R, Fischer L, Raschmann S, Schwarz J, Holzke M, Rout S, Hirschmeier C, Hamann J, Herwig U, Richter J, Baumgardt J, Weinmann S. Utilization of Psychiatric Hospital Services Following Intensive Home Treatment: A Nonrandomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2445042. doi: 10.1001/jamanetworkopen.2024.45042. PMID 39546314